CLINICAL TRIAL: NCT05488444
Title: A Feasibility and Acceptability Pilot Study Evaluating a Patient-Specific Targeted Intervention Using Patient Navigators or Routine Clinical Care
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 0 Participants Accrued
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-0150; ASCO (Other Grant/Funding Number: FP00004259); NCI-2022-06440 (Other: NCI-CTRP Clinical Trial Registry)
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Investigational Group) (Experimental): Participants will complete an in-depth patient needs checklist to identify patient-specific barriers that could lead to a delay with starting chemotherapy.
  Interventions: Behavioral: Navigator Phone Calls; Behavioral: Exit Interview
- Group 2 (Control Group) (Experimental): Participants will follow routine clinical care, where chemotherapy start date is determined by the provider and patient.
  Interventions: Behavioral: Navigator Phone Calls; Behavioral: Exit Interview

INTERVENTIONS:
Behavioral: Navigator Phone Calls — The patient navigator will call you every week as described above in "Study Groups." These phone calls will continue until you begin receiving chemotherapy.
Behavioral: Exit Interview — Participants will be asked to complete an exit interview either in person or by phone

SUMMARY:
Project Lets start will provide individual support to breast cancer patients with the goal of reducing delay to chemotherapy initiation. In this study participants will identify areas of need and work with patient navigators who will provide weekly 1-1 support throughout patient's journey to beginning chemotherapy

DETAILED DESCRIPTION:
OBJECTIVES:

Among patients with early-stage breast cancer, delays with the administration of chemotherapy significantly reduce its benefit. Interventions aimed at reducing TTC have the potential of improving outcomes and reducing health disparities. In this study we propose to develop an effective targeted intervention that is culturally sensitive and that addresses the roots of chemotherapy delay.

Our objective is to conduct a pilot study randomizing patients with breast cancer, in whom adjuvant or neoadjuvant chemotherapy has been recommended, to a culturally sensitive and patient-specific targeted intervention using patient navigators or routine clinical care

Primary Aim: To establish feasibility and acceptability.

We hypothesize that the intervention will be feasible and accepted by participants.

Secondary Aim: Explore TTC according to treatment arm. We hypothesize that the TTC will be shorter among participants randomized to the intervention

Exploratory Aim: 1) To determine if social support, interpersonal trust in a physician, and general self-efficacy changed from baseline to the end of the intervention; and 2) to determine if that change was similar between participants randomized to the intervention compared to the control arm.

We hypothesize that there will be favorable changes in scores among participants randomized to the intervention, while no change will occur among those randomized to the control arm.

ELIGIBILITY:
Inclusion Criteria:

I. At least 18 years of age. II. Diagnosis of primary invasive breast cancer. III. Chemotherapy (adjuvant or neo-adjuvant) recommended by treating physician (including pregnant women in 2nd or 3rd trimester).

IV. Patient of the University of Texas MD Anderson Cancer Center or planning on receiving treatment at our Institution.

V. Can speak, read, and understand English and/or Spanish. VI. Participant can provide consent for themself

Exclusion Criteria:

I. Hospitalized for a critical condition or who are considered medically unstable by their medical team.

II. Patients that have been previously treated with chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
General Self-Efficacy (GSE) Scale Questionnaires | through study completion and average of 1 year.
  Responses are made on a 4-point scale, ranging from 1 (not at all true) to 4 (exactly true). Scores could range from a composite score of 10 to 40, with higher score indicating more self-efficacy.25

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Chavez Mac Gregor, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT05488444/ICF_000.pdf